CLINICAL TRIAL: NCT06760429
Title: Comparative Evaluation of Pectoral Nerve Block Type II Versus Rhomboid Intercostal and Subserratus Plane Block in Breast Cancer Mastectomy for Postoperative Analgesia: a Randomized, Controlled Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Inner Mongolia Baogang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024-MER-302
Record Dates: First submitted 2025-01-03; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subserratus Plane Block (Experimental): Once the needle tip reached the fascial plane between the pectoralis minor and serratus anterior muscles and there was no blood aspiration, 15 mL of 0.375% ropivacaine was injected. Then the needle was withdrawn until the needle tip reached the fascial plane between the pectoralis major and pectoralis minor muscles, and another 15 mL of 0.375% ropivacaine was injected. After the nerve block was implemented, the area of sensory block was marked, and the spread of the local anesthetic was monitored by ultrasound. Alcohol swabs and pinprick tests were used to detect cold and pain sensations.
  Interventions: Procedure: Subserratus Plane Block
- Pectoral Nerve Block Type 2 (Experimental)
  Interventions: Procedure: Pectoral Nerve Block Type II

INTERVENTIONS:
Procedure: Pectoral Nerve Block Type II — In the PECS II group,once the needle tip reached the fascial plane between the pectoralis minor and serratus anterior muscles and there was no blood aspiration, 15 mL of 0.375% ropivacaine was injected. Then the needle was withdrawn until the needle tip reached the fascial plane between the pectoralis major and pectoralis minor muscles, and another 15 mL of 0.375% ropivacaine was injected. After the nerve block was implemented, the area of sensory block was marked, and the spread of the local anesthetic was monitored by ultrasound. Alcohol swabs and pinprick tests were used to detect cold and pain sensations.
  Arms: Pectoral Nerve Block Type 2
Procedure: Subserratus Plane Block — In the RISS group,the linear ultrasound probe was placed in the sagittal plane at the level of the 5th to 6th thoracic vertebrae (T5-6), just medial to the scapula, to identify the trapezius, rhomboid major, and intercostal muscles. A 21-gauge puncture needle was inserted in a cranial-to-caudal direction into the plane between the rhomboid major and intercostal muscles. When there was no blood aspiration, 20 mL of 0.375% ropivacaine was injected. After that, the ultrasound probe was moved caudally and laterally to identify the tissue plane between the serratus anterior and external intercostal muscles for performing the subserratus block at the level of the 8th to 9th thoracic vertebrae (T8-9). The puncture needle was advanced from the previous position, and when there was no blood aspiration again, an additional 20 mL of 0.375% ropivacaine was injected.
  Arms: Subserratus Plane Block

SUMMARY:
This study aimed to investigate the analgesic effects of Pectoral Nerve Block Type II and Rhomboid Intercostal and Subserratus Plane Block after radical mastectomy for breast cancer.This prospective, double-blind, randomized controlled trial recruited 67 female patients with complete follow-up records who underwent unilateral modified radical mastectomy (MRM) at Inner Mongolia Baotou Steel Hospital from December 1, 2023 to December 1, 2024. Subjects were assigned to the observation group and the control group at a 1:1 ratio using a random number table. Among them, 30 patients who received pectoral nerve block (PECS II) for analgesia were included in the observation group, and 30 patients who received Rhomboid Intercostal and Subserratus (RISS) block for analgesia were included in the control group. The primary outcomes included the 40-item Quality of Recovery (QoR-40) scores at 6 hours and 24 hours after surgery, and the Visual Analogue Scale (VAS) pain scores in the Post-Anesthesia Care Unit (PACU), as well as at 2 hours, 6 hours, 12 hours, 24 hours, and 48 hours after surgery.T he secondary outcomes included the consumption of sufentanil in patient-controlled intravenous analgesia (PCIA) after surgery, the number of effective compressions, the use of remifentanil during the operation, the number of additional analgesic administrations, the sleep quality on the first day after surgery, and the incidences of block-related complications and postoperative adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients met the diagnostic criteria of breast cancer;
* tolerance to surgery and anesthesia

Exclusion Criteria:

* Patients with severe systemic diseases or anesthesia problems: Such patients were excluded to ensure safety and avoid the occurrence of irrelevant complications;
* Those with coagulation disorders;
* Patients with puncture contraindications or infections;
* Those allergic to local anesthetics;
* Those who refused to sign the informed consent form;
* Patients with cognitive or communication problems

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale | From PACU entry to 48 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No